CLINICAL TRIAL: NCT06273709
Title: The Value of Visual Inspection When Remotely Diagnosing Basal Cell Carcinoma on Optical Coherence Tomography Scans: a Diagnostic Case-control Study
Brief Title: Remote Assessment of OCT Scans for BCC Detection
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-3698
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Optical coherence tomography; Imaging; Non-melanoma skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCT scans without clinical/dermoscopic photographs: OCT scans will be used from a pre-existing registry. The OCT scans are made of lesions clinically suspect for BCC. All patients underwent punch biopsy conform regular care.
  Interventions: Device: Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner
- OCT scans with clinical/dermoscopic photographs: The same OCT scans will be used . OCT assessment is performed in conjunction with clinical and dermoscopic photographs.
  Interventions: Device: Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner

INTERVENTIONS:
Device: Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner — (Michelson Diagnostics Maidstone, Kent, UK; resolution <7.5 µm lateral, <5 µm axial; depth of focus 1.0 mm; scan area 6 × 6 mm).

SUMMARY:
Basal cell carcinoma (BCC) is the most common form of cancer and entails approximately 80% of all cutaneous malignancies. This locally destructive neoplasm is commonly diagnosed by punch biopsy which is considered painful, causes procedural scarring and carries a small risk of infection and re-bleeding associated with invasive procedures. Moreover, awaiting the results of the subsequent histopathological examination causes treatment delay and can be stressful for the patient. The drawbacks of biopsy could be overcome by optical coherence tomography (OCT), a non-invasive diagnostic modality that may replace biopsy in up to 66% of patients. However, OCT assessors are scarce which hinders the implementation of OCT. This problem may be addressed by teledermatology in which remote OCT assessment by an assessor facilitates simultaneous assessment for multiple clinics. Remote OCT assessment withholds the OCT assessor from visually inspecting the lesion. But the effect of visual inspection on the diagnostic accuracy remains unknown and the question arises whether visual inspection is necessary for accurate OCT assessment. In this diagnostic case-control study we will determine whether distant OCT assessment without visual information on the lesion is non-inferior to distant OCT assessment with clinical and dermoscopic photographs (CDP-OCT).

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Underwent OCT scan and punch biopsy for lesions suspect for BCC

Exclusion Criteria:

* Unable to sign informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Included cases contain OCT scans of patients with lesions suspect for BCC. Three OCT assessors will be included in this study to assess the OCT scans with and without clinical and dermoscopic photographs.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of high-confidence BCC diagnosis with and without clinical/dermoscopic photographs | Measured before December 31st 2024
  Diagnostic accuracy of a high confidence diagnosis (confidence-score 4) will be expressed by diagnostic parameters, such as sensitivity, specificity, positive predictive value (PPV), negative predicitive value (NPV), and diagnostic odds ratios (DOR) with 95% confidence intervals. The primary outcome in this study is specificity of a high confidence diagnosis, defined as the proportion of histological non-BCC lesions that are classified as non-BCC on OCT.

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon reasonable request.

REFERENCES:
- [Derived] Wolswijk T, Nelemans PJ, van Leersum F, Cruts E, Gerarda Moermans MM, Vreven L, Hillen LM, Mosterd K. The Impact of Clinical and Dermoscopic Photographs on the Diagnostic Accuracy of Remote Optical Coherence Tomography Assessment for Basal Cell Carcinoma Detection: A Comparative Diagnostic Study. Int J Dermatol. 2025 Dec 10. doi: 10.1111/ijd.70189. Online ahead of print. PMID 41373084